CLINICAL TRIAL: NCT06548789
Title: Neoadjuvant Immune Checkpoint Blockade + a Prebiotic Food-enriched Dietary Intervention to Optimize Immune Response in Melanoma: NEO-PreFED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0388; NCI-2024-06747 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prebiotic food-enriched diet (PreFED) (Experimental): Participants will identified from the clinic schedules and/or referred from participant's treating oncologists.
  Interventions: Dietary Supplement: Prebiotic Xnack Packouts

INTERVENTIONS:
Dietary Supplement: Prebiotic Xnack Packouts — Prebiotic snack packouts (distributed every two weeks) and diet counseling to support increased consumption of prebiotic foods which provide dietary fiber, plant-based protein and other nutrients selectively fermented by the microbiome (e.g., pulses and legumes).

SUMMARY:
To Determine the feasibility, compliance and adherence to PreFED intervention in resectable melanoma patients initiating neoadjuvant Ipi/Nivo.

DETAILED DESCRIPTION:
Primary Objectives:

Determine the feasibility, compliance and adherence to PreFED intervention in patients with resectable melanoma initiating neoadjuvant combination ICB therapy.

Secondary Objectives:

1. Determine the safety (AEs) and tolerability (GSRS-IBS) of the dietary intervention during the neoadjuvant phase and maintenance phases
2. Assess the rate of immune related adverse events in patients of dietary intervention + ICB during neoadjuvant and maintenance phases.
3. Determine the objective response rate (ORR) to dietary intervention + ICB as determined by RECIST1.1 after 2 cycles of neoadjuvant ICB + diet
4. Determine the pathological response rate (pRR) to neoadjuvant ICB + dietary intervention
5. Determine the Event-free Survival (EFS), Relapse-free Survival (RFS), and Overall Survival (OS) to neoadjuvant ICB + dietary intervention

Exploratory Objectives:

1. Assess the effect of dietary intervention + ICB on gut microbiome composition at completion of neoadjuvant phase and maintenance phase
2. Assess the effects of dietary intervention + neoadjuvant ICB on gut metabolic output and systemic metabolism at completion of neoadjuvant phase and maintenance phase
3. Assess the effects of dietary intervention + neoadjuvant ICB on systemic and tumor immunity at time of surgery
4. Assess the effects of dietary intervention + neoadjuvant ICB on quality of life and other patient reported outcomes (PROs) during neoadjuvant and maintenance phases

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Body mass index (BMI) 18.5-45 kg/m2
3. Able to self-complete study assessments monitoring diet and gastrointestinal symptom burden
4. ECOG performance status of 0 or 1
5. Histologically confirmed resectable stage IIIB-D or oligometastatic Stage IV cutaneous melanoma or locally invasive/advanced mucosal melanoma as determined by multidisciplinary review
6. Planned initiation of standard-of-care neoadjuvant ipilimumab +/- nivolumab or nivolumab +/- relatlimab
7. Measurable disease per RECIST 1.1
8. WOCP must have negative UPT within 1 week of beginning dietary intervention.
9. Self-reported willingness to eat the provided foods (with some tailoring to their food preferences)
10. Self-reported willingness to comply with scheduled visits, undergo venipuncture, provide stool samples.
11. Archival tissue specimen or planned to undergo tumor biopsy as part of standard of care treatment.

Exclusion Criteria:

1. Uveal melanoma
2. History of inflammatory bowel disease, total colectomy, or bariatric surgery
3. Currently taking steroids > prednisone 10 mg/day or equivalent
4. Medical contraindications to the intervention diet as determined by the treating physician
5. Self-reported major dietary restrictions, including but not limited to relevant food allergies, celiac disease, or diets such as vegan, ketogenic, extended fasting
6. Insulin-dependent diabetes or conditions requiring bile-acid sequestrants
7. Unable or unwilling to undergo study procedures
8. Intravenous (IV) antibiotic >1 dose in the past month or 1 dose IV/oral antibiotic use in past 2 weeks
9. Regularly taking supplements containing prebiotics, fiber and/or probiotics, and unable/unwilling to discontinue for the purpose of the study
10. Current smoker or heavy drinker (defined as >14 drinks per week) or current illicit drug use
11. Currently pregnant, planning to become pregnant, or lactating
12. Concurrent malignancy requiring systemic therapy other than hormonal therapy
13. Cognitively impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
The completion rate, compliance and adherence. | Up to 2 years
  The completion rate is defined as proportion of participants completed the intervention. Among subjects that complete the PreFED intervention, compliance is defined as the proportion (%) of prebiotic snacks consumed versus provided and proportion (%) of counselling sessions attended, while adherence is defined as the number of servings of prebiotic foods the participant consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Baruch, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org